CLINICAL TRIAL: NCT03743727
Title: The Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed-Dose Combination for Treatment of Egyptian Children and Adolescents With Chronic Hepatitis C (HCV)-Genotype 4
Brief Title: Treatment of Egyptian Hepatitis C Genotype 4 Infected Children and Adolescents With Combined Ledipasvir/Sofosbuvir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yassin Abdelghaffar Charity Center for Liver Disease and Research (Other)
Responsible Party: Principal Investigator, Dr. Tawhida Yassin Abdel Ghaffar, Professor, Yassin Abdelghaffar Charity Center for Liver Disease and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDV SOF T 2018
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Hepatitis C Genotype 4
MeSH Terms: interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Therapy LDV and SOF (Experimental)
  Interventions: Drug: Combined therapy LDV and SOF

INTERVENTIONS:
Drug: Combined therapy LDV and SOF — All patients will receive ledipasvir/sofosbuvir fixed dose combination for 12 weeks. Patients weighing 35 kg or more will receive the adult dose: ledipasvir (90 mg)/sofosbuvir (400 mg). Patients weighing below 35 kg will receive half the adult dose: ledipasvir (45 mg)/sofosbuvir (200 mg).
  Other Names: ledipasvir and sofosbuvir

SUMMARY:
This is an open, uncontrolled study of twenty-five chronic HCV infected patients carried out at Yassin Abdel Ghaffar Charity Center for Liver Disease and Research. The aim of this study is to investigate the safety & efficacy of combined therapy ledipasvir (LDV) and sofosbuvir (SOF) for treating HCV Genotype 4 in children aged 8 to 18. Due to previous positive results in other clinical studies of this drug it is expected that the drug will have high safety and high efficacy. Safety will be measured by checking for adverse effects, while efficacy will be measured by Real-Time Quantitative Polymerase Chain Reaction (qPCR) detecting viral nucleic acids in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* HCV chronic infection
* Treatment naive and treatment experienced (previous interferon treatment)
* No cirrhosis or compensated cirrhosis

Exclusion Criteria:

* Co-infection with Hepatitis B (HBV)
* Other associated chronic liver illness
* Patients with history of hematemesis (non-cirrhotic portal hypertension)
* Patients with decompensated cirrhosis (as indicated by biopsy, fibroscan)
* Patients on drugs known to interact unfavorably (Amioidarone, ..)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | During the 12 weeks of treatment.
  The presence of any adverse effects will be used to characterize this outcome measure.
Sustained Viral Clearance | At Week 12 after end of treatment.
  HCV RNA qPCR will be used to determine if the target of viral clearance has been established. Detection limit of the kit is 12 IU/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Tawhida Y. Abdel Ghaffar, MD, Principal Investigator — Yassin Abdel Ghaffar Charity Center for Liver Disease and Research
Locations (1):
- Professor Yassin Abdel Ghaffar Charity Center for Liver Disease and Research, Madīnat an Naşr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No